CLINICAL TRIAL: NCT02049762
Title: Aspirin Impact on Platelet Reactivity in Acute Coronary Syndrome Patients on Novel P2Y12 Inhibitors Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Shlomi Matetzky, Head of The Cardiac Intensive Care Unit, Sheba Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 0813-13-SMC
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Acute Coronary Syndrome; Platelet Function and Reactivity Tests; Novel P2Y12 Inhibitors
Keywords: novel P2Y12 inhibitors; aspirin; platelet reactivity; acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- P2Y12 inhibitors and aspirin (Active Comparator): ACS patients on novel P2Y12 inhibitors and aspirin
  Interventions: Drug: Aspirin
- P2Y12 inhibitors and placebo (Placebo Comparator): ACS patients on novel P2Y12 inhibitors and placebo
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Aspirin 100 mg vs. placebo in ACS patients on P2Y12 inhibitors a month following PCI.

SUMMARY:
Thus far, no study has evaluated the impact on aspirin in addition to the newer and more potent P2Y12 inhibitors, among ACS patients and current guidelines recommend dual anti-platelet therapy consisting of aspirin and a novel P2Y12 inhibitor in this population.

Objective The investigators goal is to examine the effect of aspirin in addition to new anti-platelet agent (ticagrelor\prasugrel) on platelet reactivity in comparison with placebo, among ACS patients treated percutaneously.

Design The proposed study is a randomized-controlled, double blind trial, conducted among ACS patients treated percutaneously. Eligible patients will recruited during hospitalization due to ACS after percutaneous coronary intervention (PCI), and randomization by envelopes on 1:1 basis will take place a month after the index event, at a follow-up visit at the cardiac clinic.

Platelet function and Endothelial function tests will be taken a month after the index event, and at a 2 weeks periods following aspirin/placebo therapy, cross-over and return to open-label aspirin.

End-points platelet function tests will be compared between aspirin and placebo therapy and before and after the cross-over.

DETAILED DESCRIPTION:
Introduction:

Current knowledge and data support the use of dual anti-platelets for patients after acute coronary syndrome (ACS). Novel P2Y12 inhibitors have shown their superiority on clopidogrel in regarding morbidity and mortality, but at the cost of higher bleeding rates - even in lower doses of aspirin there is increase risk for gastrointestinal (GI) bleeding. In a geographical analysis of the PLATO trial it has been shown difference at outcome. When higher dose of aspirin were used, the superiority of ticagrelor was reduced.

The use of platelet reactivity tests have been proved and acknowledged in their usefulness for gauging bleeding and ischemic risks. Few studies have shown that clopidogral is inhibiting not only the ADP activity, but also the arachidonic acid (AA) pathway that is considered aspirin specific pathway. Examining the effect of potent P2Y12 inhibitors in healthy volunteers have shown increased inhibition of the AA pathway. Not only that the adding of aspirin, have shown little effect on inhibition of AA pathway.

It has been demonstrated that vascular endothelial function is inversely correlated to platelet reactivity in both individuals without established cardiovascular disease (controls) and acute myocardial infarction patients.

Objective Our goal is to examine the effect (platelet function test and endothelial function) of aspirin while added to novel P2Y12 inhibitors treated ACS patients.

Design The proposed study is a randomized-controlled, double blind trial, conducted among ACS patients treated percutaneously. Eligible patients will recruited during hospitalization due to ACS after percutaneous coronary intervention (PCI), and randomization by envelopes on 1:1 basis will take place a month after the index event, at a follow-up visit at the cardiac clinic.

Platelet function and Endothelial function tests will be taken a month after the index event, and at a 2 weeks periods following aspirin/placebo therapy, cross-over and return to open-label aspirin.

Study end-points The primary end-point is platelet function tests in response to AA. Secondary end-points will include endothelial function and platelet reactivity according to the platelet activity and VerifyNow test in response to ADP and platelet activation Clinical outcomes including all-cause and cardiac mortality and hospitalizations, recurrent ischemia and stent thrombosis, and bleeding events along with blood transfusions, will be recorded as safety end-points.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* ACS defined according to the 3rd universal definition of MI
* PCI therapy

Exclusion Criteria:

* Indication for anticoagulant therapy
* ACS on new P2Y12 inhibitors treatment
* Contraindication to P2Y12 therapy
* Renal failure defined as creatinine ≥1.5 mg/dL
* Non-compliance
* Life-threatening extra-cardiac disease or malignancy with a life expectancy below 1 year
* Inability to sign an informed consent
* Participation in another trial during the previous 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity | one month
  platelet reactivity in response to arachidonic acid

SECONDARY OUTCOMES:
platelet reactivity | one month
  platelet reactivity in response to ADP

OTHER OUTCOMES:
clinical outcome | two months
  hospitalizations and mortality

CONTACTS AND LOCATIONS:
Overall Officials: Shlomi Matezky, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Background] Wiviott SD, Braunwald E, McCabe CH, Montalescot G, Ruzyllo W, Gottlieb S, Neumann FJ, Ardissino D, De Servi S, Murphy SA, Riesmeyer J, Weerakkody G, Gibson CM, Antman EM; TRITON-TIMI 38 Investigators. Prasugrel versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2007 Nov 15;357(20):2001-15. doi: 10.1056/NEJMoa0706482. Epub 2007 Nov 4. PMID 17982182
- [Background] Yusuf S, Zhao F, Mehta SR, Chrolavicius S, Tognoni G, Fox KK; Clopidogrel in Unstable Angina to Prevent Recurrent Events Trial Investigators. Effects of clopidogrel in addition to aspirin in patients with acute coronary syndromes without ST-segment elevation. N Engl J Med. 2001 Aug 16;345(7):494-502. doi: 10.1056/NEJMoa010746. PMID 11519503
- [Background] Mahaffey KW, Wojdyla DM, Carroll K, Becker RC, Storey RF, Angiolillo DJ, Held C, Cannon CP, James S, Pieper KS, Horrow J, Harrington RA, Wallentin L; PLATO Investigators. Ticagrelor compared with clopidogrel by geographic region in the Platelet Inhibition and Patient Outcomes (PLATO) trial. Circulation. 2011 Aug 2;124(5):544-54. doi: 10.1161/CIRCULATIONAHA.111.047498. Epub 2011 Jun 27. PMID 21709065
- [Background] Tantry US, Bonello L, Aradi D, Price MJ, Jeong YH, Angiolillo DJ, Stone GW, Curzen N, Geisler T, Ten Berg J, Kirtane A, Siller-Matula J, Mahla E, Becker RC, Bhatt DL, Waksman R, Rao SV, Alexopoulos D, Marcucci R, Reny JL, Trenk D, Sibbing D, Gurbel PA; Working Group on On-Treatment Platelet Reactivity. Consensus and update on the definition of on-treatment platelet reactivity to adenosine diphosphate associated with ischemia and bleeding. J Am Coll Cardiol. 2013 Dec 17;62(24):2261-73. doi: 10.1016/j.jacc.2013.07.101. Epub 2013 Sep 27. PMID 24076493
- [Background] Hobson AR, Qureshi Z, Banks P, Curzen NP. Effects of clopidogrel on "aspirin specific" pathways of platelet inhibition. Platelets. 2009 Sep;20(6):386-90. doi: 10.1080/09537100903003227. PMID 19811222
- [Background] Armstrong PC, Dhanji AR, Tucker AT, Mitchell JA, Warner TD. Reduction of platelet thromboxane A2 production ex vivo and in vivo by clopidogrel therapy. J Thromb Haemost. 2010 Mar;8(3):613-5. doi: 10.1111/j.1538-7836.2009.03714.x. Epub 2009 Dec 3. No abstract available. PMID 19995405
- [Background] Armstrong PC, Leadbeater PD, Chan MV, Kirkby NS, Jakubowski JA, Mitchell JA, Warner TD. In the presence of strong P2Y12 receptor blockade, aspirin provides little additional inhibition of platelet aggregation. J Thromb Haemost. 2011 Mar;9(3):552-61. doi: 10.1111/j.1538-7836.2010.04160.x. PMID 21143373
- [Background] Kirkby NS, Leadbeater PD, Chan MV, Nylander S, Mitchell JA, Warner TD. Antiplatelet effects of aspirin vary with level of P2Y(1)(2) receptor blockade supplied by either ticagrelor or prasugrel. J Thromb Haemost. 2011 Oct;9(10):2103-5. doi: 10.1111/j.1538-7836.2011.04453.x. No abstract available. PMID 21812912
- [Background] Warner TD, Armstrong PC, Curzen NP, Mitchell JA. Dual antiplatelet therapy in cardiovascular disease: does aspirin increase clinical risk in the presence of potent P2Y12 receptor antagonists? Heart. 2010 Nov;96(21):1693-4. doi: 10.1136/hrt.2010.205724. PMID 20956485
- [Background] Lanas A, Garcia-Rodriguez LA, Arroyo MT, Gomollon F, Feu F, Gonzalez-Perez A, Zapata E, Bastida G, Rodrigo L, Santolaria S, Guell M, de Argila CM, Quintero E, Borda F, Pique JM; Asociacion Espanola de Gastroenterologia. Risk of upper gastrointestinal ulcer bleeding associated with selective cyclo-oxygenase-2 inhibitors, traditional non-aspirin non-steroidal anti-inflammatory drugs, aspirin and combinations. Gut. 2006 Dec;55(12):1731-8. doi: 10.1136/gut.2005.080754. Epub 2006 May 10. PMID 16687434
- [Background] Hallas J, Dall M, Andries A, Andersen BS, Aalykke C, Hansen JM, Andersen M, Lassen AT. Use of single and combined antithrombotic therapy and risk of serious upper gastrointestinal bleeding: population based case-control study. BMJ. 2006 Oct 7;333(7571):726. doi: 10.1136/bmj.38947.697558.AE. Epub 2006 Sep 19. PMID 16984924
- [Background] Wang TY, Xiao L, Alexander KP, Rao SV, Kosiborod MN, Rumsfeld JS, Spertus JA, Peterson ED. Antiplatelet therapy use after discharge among acute myocardial infarction patients with in-hospital bleeding. Circulation. 2008 Nov 18;118(21):2139-45. doi: 10.1161/CIRCULATIONAHA.108.787143. Epub 2008 Nov 3. PMID 18981304
- [Background] Roy P, Bonello L, Torguson R, de Labriolle A, Lemesle G, Slottow TL, Steinberg DH, Kaneshige K, Xue Z, Satler LF, Kent KM, Suddath WO, Pichard AD, Lindsay J, Waksman R. Impact of "nuisance" bleeding on clopidogrel compliance in patients undergoing intracoronary drug-eluting stent implantation. Am J Cardiol. 2008 Dec 15;102(12):1614-7. doi: 10.1016/j.amjcard.2008.07.063. Epub 2008 Sep 27. PMID 19064014